CLINICAL TRIAL: NCT02842944
Title: Weaning From Mechanical Ventilation Comparison of Open-loop Decision Support System and Routine Care
Acronym: BEACON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI2016_843_0018
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open loop weaning group (Beacon) (Experimental): mechanical ventilation following advice from the Beacon Caresystem
  Interventions: Device: open loop weaning group (Beacon)
- Routine care (Active Comparator): * Connect and start Beacon with advice disabled
  * Standardized routine care
  Interventions: Other: Routine care

INTERVENTIONS:
Device: open loop weaning group (Beacon) — mechanical ventilation following advice from the Beacon Caresystem
  Arms: open loop weaning group (Beacon)
Other: Routine care — Standardized routine care
  Arms: Routine care

SUMMARY:
The purpose of this study is to compare mechanical ventilation following advice from the Beacon Caresystem to that of routine care in patients from the state of requiring invasive mechanical ventilation until successful extubation. The Beacon Caresystem will be compared to routine care to investigate whether use of the system results in similar care and reduced time for weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is on invasive mechanical ventilation more 48 hours
* Age > 18 years
* Patients are ventilated using Maquet Servo-I, Draeger Infinity V500 or Draeger Evita XL mechanical ventilators in "pressure support", "volume controlled", or "pressure controlled" ventilation modes.
* Haemodynamically stable (mean blood pressure ≥ 65 mmHg)
* Patients or, in the case that the patient is unable, next of kin understand and accept oral and written information describing the study or patient consent retrospectively in case of emergency inclusion.

Exclusion Criteria:

* The absence of an arterial catheter for blood sampling.
* Medical history of home mechanical ventilation
* Severe ARDS (PaO2/FiO2 ≤ 100 mmHg)
* Head trauma or other conditions where intra-cranial pressure may be elevated and tight regulation of arterial CO2 level is paramount.
* Severe neurological patients (Glasgow coma score <10, neurologic damage with limited prognosis, stroke hemiplegia).
* Known or suspected severe myopathy or neuropathy (including ICU neuromyopathy)
* Quadriplegia
* Severe heart failure
* Broncho alveolar fistula with more than 100ml leakage
* History of home mechanical ventilation
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 14 days
  time from initial intubation and until successful extubation, with successful extubation defined as ≥ 7 days of unassisted spontaneous breathing after extubation.
Time to successful extubation | Successful extubation is defined as ≥ 7 days of unassisted spontaneous breathing after extubation
  time from randomization and until successful extubation.
Time from support mode to successful extubation | 14 days
  the time after point of randomization, from initiation of support modes of ventilation and until successful extubation

CONTACTS AND LOCATIONS:
Overall Officials: Elie ZOGHEIB, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France